CLINICAL TRIAL: NCT03817788
Title: Randomized Controlled Trail of Polyethylene Glycol vs Sodium Phosphate for Colonic Cleansing of Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong Yang (Other)
Collaborators: Xu Hong (Unknown)
Responsible Party: Sponsor-Investigator, Dong Yang, Doctor, Jilin University
Organization: Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 130022
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Polyethylene Glycol; Sodium Phosphate
MeSH Terms: interventions — Polyethylene Glycols; sodium phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyethylene glycol group (group P) (Active Comparator): For all patients of this group, polyethylene glycol solution should be taken orally for colonic cleansing of colonoscopy
  Interventions: Drug: polyethylene glycol
- sodium phosphate group (group S) (Experimental): For all patients of this group, sodium phosphate solution should be taken orally for colonic cleansing of colonoscopy
  Interventions: Drug: sodium phosphate

INTERVENTIONS:
Drug: polyethylene glycol — All patients should receive dietary guidance, and eat a low-residue diet three days before colonoscopy. For polyethylene glycol group (group P): the day before colonoscopy, 750 mL (1 box) of polyethylene glycol solution should be drunk 2 hours after dinner; the other 1500 ml (2 boxes) of polyethylene glycol solution should be taken 4-6 hours before the examination. After oral laxatives were finished, 20 ml dimethicone would be taken orally as defoamer. All the enteroscopy should by performed by the same juniar clinician, and related indicators were recorded.
  Arms: polyethylene glycol group (group P)
Drug: sodium phosphate — All patients should receive dietary guidance, and eat a low-residue diet three days before colonoscopy. For sodium phosphate group (group S), 750 mL (1 box) of sodium phosphate solution should be drunk 2 hours after dinner; and the other 750 mL (1 box) of sodium phosphate solution should be taken 4-6 hours before the examination. After oral laxatives were finished, 20 ml dimethicone would be taken orally as defoamer. All the enteroscopy should by performed by the same clinician, and related indicators were recorded.
  Arms: sodium phosphate group (group S)

SUMMARY:
This study is to compare polyethylene glycol and sodium phosphate for colonic cleansing of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients meet the following criteria: 1) age 18-60 years; 2) BMI 18.9-28; 3) Heart, lung, liver, and kidney function can tolerate colonoscopy; 4) Patients and their families are able to understand and be willing to participate in this clinical study and to sign informed consent

Exclusion Criteria:

* 1) colorectal surgery history (except appendectomy); 2) patients with intestinal obstruction, incomplete obstruction, intestinal hemorrhage; 3) patients with renal insufficiency; 4) patients with hirschsprung disease; 5) patients with inflammatory bowel disease during active period, which affects intestinal observation; 6) patients who are bedridden and lose the moving ability ; 7) have a history of severe mental illness; 8) pregnant or lactating women; 9) patients with other clinical conditions considered by some researchers should not participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 586 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Cleansing quality | during the procedure of colonoscopy
  The quality of colon cleansing was assessed by the endoscopist with Boston bowel preparation scale.

SECONDARY OUTCOMES:
the duration of the procedure | during the procedure of colonoscopy
  time to cecal intubation and withdrawal time
patient tolerance | before the procedure of colonoscopy
  patient tolerance about oral laxatives.
the degree of difficulty of the procedure | at the end of the procedure of colonoscopy
  6-point scale: extremely easy, easy, fairly easy, fairly difficult, difficult, extremely difficult
polyps or other endoscopic lesions | at the end of the procedure of colonoscopy
  For polyps or other endoscopic lesions, a histopathologic diagnosis was systematically obtained and recorded
patient pain | at the end of the procedure of colonoscopy
  (visual analog scale, 0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.